CLINICAL TRIAL: NCT03704090
Title: Non-pharmacological Prevention of Postoperative Delirium by Occupational Therapy Teams in Patients Older Than 75 Years Undergoing High-risk Elective Surgery
Brief Title: Non-pharmacological Prevention of Postoperative Delirium by Occupational Therapy Teams
Acronym: PREPODOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Hospital de San Jose (Other); Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Antonello Penna, Anesthesiologist, Assistent Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SA17I0030
Record Dates: First submitted 2018-10-07; First posted 2018-10-12 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Delirium; Aging Disorder
Keywords: Postoperative Delirium; Prevention Measure; Non-pharmacological; Subsyndromal Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: Elderly patients who will undergo major surgery will be randomized to 2 prevention groups of postoperative delirium:
  1. Control: standard non-pharmacological prevention measures for 5 days after surgery.
  2. Intervention: occupational therapist plus standard non-pharmacological prevention measures for 5 days after surgery.
Who Masked: Care Provider, Investigator
Masking Description: Patients were randomized in 16 blocks of 10 patients and only one investigator has the randomized information. This researcher will not have any role in the recruitment, intervention, and diagnosis of postoperative delirium. Also, the analysis of data will be performed by researchers who will be masked to the randomization information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard non-pharmacological intervention during 5 days after surgery.
  Interventions: Behavioral: Standard non-pharmacological prevention intervention
- Treatment (Experimental): Occupational therapy intervention twice a day plus standard non-pharmacological prevention intervention during 5 days after surgery.
  Interventions: Behavioral: Occupational therapy intervention; Behavioral: Standard non-pharmacological prevention intervention

INTERVENTIONS:
Behavioral: Occupational therapy intervention — Prevention of postoperative delirium by occupational therapy intervention
  Arms: Treatment
Behavioral: Standard non-pharmacological prevention intervention — Prevention of postoperative delirium using standard non-pharmacological prevention measures

SUMMARY:
In the world, 230 million surgeries are performed every year and US data indicates that more than a third of patients who undergo surgery are older than 65 years, in which between 10 and 70% develop postoperative delirium (POD). Patients who develop POD have poor outcomes, such as a longer hospital stay, a deterioration in functional and cognitive status, high mortality rates, and an increase in health costs.

Delirium is an entity that in a significant percentage is preventable, thus preventing the development of POD is fundamental. In fact, in older adults hospitalized in the no surgical ward, the implementation of non-pharmacological prevention measures of delirium has consistently shown to significantly prevent the development of this condition. However, limited information is available about the usefulness of non-pharmacological intervention protocols applied in the perioperative context to prevent POD.

The main aim of this project is to determine whether the application of non-pharmacological measures during the perioperative period prevents POD in elderly patients undergoing highly complex elective surgeries.

The hypothesis is that the application of these measures decreases the incidence of delirium in this population.

DETAILED DESCRIPTION:
To determine whether non-pharmacological measures decrease the incidence of POD during the perioperative period in elderly patients undergoing highly complex elective surgeries, it will be performed a randomized clinical trial, where two groups of patients older than 75 years undergoing highly complex elective surgeries will be compared:

1. The first group will receive a protocol of non-pharmacological interventions implemented by occupational therapy teams to prevent delirium plus standard non-pharmacological prevention interventions.
2. The second group will only receive standard non-pharmacological prevention interventions.

This study will be carried out in the surgical units of the Hospital Clinico de la Universidad de Chile (HCUCH) and in the Hospital San Jose (HSJ).

The expected result is to demonstrate that the interventions carried out by occupational therapists decrease the incidence of DPO in a significant way in comparison with standard prevention intervention.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission for highly complex elective surgery

Exclusion Criteria:

* History of cognitive impairment.
* A low score in Mini-Mental State Examination (MMSE): <23 points if the patient has 6 or more years of schooling, and <18 points if the patient has <6 years of schooling.
* Severe communication disorder and cultural language limitation (language other than Spanish).
* Delirium on admission or prior to the start of the intervention (measured with CAM).
* Patient enrolled in another study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Delirium | 5 days
  Developing postoperative delirium evaluated by CAM (complete criteria for delirium diagnostic)
Subsyndromal delirium | 5 days
  Developing postoperative subsyndromal delirium evaluated by CAM (incomplete criteria for delium diagnostic)

SECONDARY OUTCOMES:
Lenght of hospital stay | 30 days
  Number of days between admission and discharge to the hospital
Mortality | 30 days
  Percentage of patients who die between the day of surgery and 30 days after surgery
Severity of delirium | 5 days
  Severity of delirium will be evaluated with questionnaire CAM-S
Duration of delirium | 5 days
  Number of days in which the patients have delirium

CONTACTS AND LOCATIONS:
Overall Officials: Antonello Penna, MD/PhD, Principal Investigator — University of Chile; Evelyn Alvarez, TO/MSc, Principal Investigator — Universidad Central/Universidad de Chile; Constanza Briceño, TO/MSc, Principal Investigator — University of Chile; Eduardo Tobar, MD, Principal Investigator — University of Chile; Felipe Salech, MD/PhD, Principal Investigator — University of Chile; Daniela Ponce, Ing, Principal Investigator — University of Chile; Veronica Rojas, Nurse/MSc, Principal Investigator — University of Chile; Gonzalo Navarrete, MD, Principal Investigator — University of Chile
Locations (1):
- Centro de Investigación Cínica Avanzada (CICA), Hospital Clinico de la Universidad de Chile, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alvarez EA, Garrido MA, Tobar EA, Prieto SA, Vergara SO, Briceno CD, Gonzalez FJ. Occupational therapy for delirium management in elderly patients without mechanical ventilation in an intensive care unit: A pilot randomized clinical trial. J Crit Care. 2017 Feb;37:85-90. doi: 10.1016/j.jcrc.2016.09.002. Epub 2016 Sep 10. PMID 27660922
- [Derived] Alvarez EA, Rojas VA, Caipo LI, Galaz MM, Ponce DP, Gutierrez RG, Salech F, Tobar E, Reyes FI, Vergara RC, Egana JI, Briceno CA, Penna A. Non-pharmacological prevention of postoperative delirium by occupational therapy teams: A randomized clinical trial. Front Med (Lausanne). 2023 Feb 2;10:1099594. doi: 10.3389/fmed.2023.1099594. eCollection 2023. PMID 36817762